CLINICAL TRIAL: NCT05450848
Title: A Randomised Comparison of StrataXRT to Standard Clinical Practice in the Prevention and Treatment of Radiation Dermatitis
Brief Title: StrataXRT vs. Standard Clinical Practice in the Prevention and Treatment of Radiation Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stratpharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPASX01AU002
Record Dates: First submitted 2022-06-22; First posted 2022-07-11 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Site investigators will load the digital photographs taken at each weekly assessment into each participant's MOSAIQ record. They will then send de-identified copies to the Central Trial Coordinator who will distribute them to the study investigators who will be performing the blinded assessment. Each weekly photograph will be independently assessed by two study investigators using the CTCAE 4.0 scale for radiation dermatitis (Appendix 1). The study investigators will complete the supplied photograph assessment form and return them to the Central Trial Coordinator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- StrataXRT (Experimental): Patients allocated to receive StrataXRT will be provided with StrataXRT gel to apply twice daily to the irradiated area until any radiation dermatitis that may occur has resolved. In case the patient develops radiation dermatitis that results in moist desquamation, IntraSiteTM gel (Smith and Nephew, UK) and secondary dressings will be provided.
  Interventions: Device: StrataXRT
- Standard of care (Active Comparator): Patients allocated to receive standard care will be provided with aqueous cream to apply daily to the irradiated area until any radiation dermatitis that may occur has resolved. In case the patient develops radiation dermatitis that results in moist desquamation, IntraSiteTM gel (Smith and Nephew, UK) and secondary dressings will be provided.
  Interventions: Other: Sorbolene

INTERVENTIONS:
Device: StrataXRT — StrataXRT is a flexible wound dressing for the prevention and treatment of radiation dermatitis. It is in the form of a gel which, when applied, creates a protective film that maintains skin integrity. The product is used to relieve low grade inflammatory radiation changes such as dry, itching, flaking, peeling and irritated skin. For more severe inflammatory changes with open wound components, StrataXRT reduces pain, redness and heat and helps soothe the exposed skin areas. StrataXRT can be applied where skin integrity has been compromised and may also be used in conjunction with other adjunctive treatments to improve overall results. StrataXRT contains Polydimethylsiloxanes, Siloxanes and Alkylmethyl Silicones and is transparent and odourless. It does not contain alcohols, parabens or fragrances. StrataXRT can be used with or without a secondary protective dressing. It is suitable for children and people with sensitive skin.
  Arms: StrataXRT
Other: Sorbolene — Aqueous cream (moisturizer) that soothes itchiness and dryness of the skin, and aids skin hydration. It is non-greasy, fragrance free, colour free, GMO free, paraben free and pH balanced.
  Arms: Standard of care

SUMMARY:
Current clinical practice for preventing and treating radiation dermatitis across Queensland (QLD) Health Radiation Oncology departments involves the application of aqueous cream daily to the skin of the treatment site, commencing from Day 1 of EBRT. The primary aim of this study is to assess the efficacy of StrataXRT when compared to current clinical practice in preventing and managing radiation dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer undergoing a curative course of radiation therapy using standard protocols to the following cancer sites:

  * Head and neck cancers receiving >= 60Gy who are not receiving concurrent Cetuximab
  * Intact breast receiving >= 40Gy (includes patients receiving boost fields using photon or elections)
  * Post-mastectomy chest wall (breast cancer diagnosis only) receiving >= 50Gy
  * Gynaecological cancers requiring whole pelvis irradiation receiving >= 45Gy
  * Skin cancers to the axilla/groin regions receiving >= 40Gy
* Male and female patients >18 years of age
* Patients who do not have a known allergy to silicon
* Patients who are able to attend the four post-treatment weekly skin assessment appointments

Exclusion Criteria:

Ineligible participants are patients undergoing a course of curative radiation therapy:

* Who are participating in another interventional study
* With an allergy to product content (standard or StrataXRT)
* With an existing skin rash, ulceration or open wound in the treatment area
* With a pre-existing systemic skin disease (dermatological conditions, connective tissue disorders)
* Who have had previous radiation therapy to the current treatment area
* Who are on immuno-suppression drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | From radiotherapy start, until to 4 weeks post radiation therapy; up to 3 months
  Radiation dermatitis reaction as assessed by blinded assessment of digital photographs using the CTCAE v4.0 radiation dermatitis grades. CTCAE v4.0 severity grades are categorical with 5 possible categories (1, 2, 3, 4, 5). Grade 1 represents the weakest form of radiation dermatitis. Higher CTCAE Grades represent increasing radiation dermatitis severity.
Radiation induced skin reaction assessment scale (RISRAS) | From radiotherapy start, until to 4 weeks post radiation therapy; up to 3 months
  Radiation dermatitis reaction as assessed by the clinician during patient consultations using the eviQ RISRAS form. RISRAS scale is continuous scale from 0 to 36, with higher RISRAS scores representing higher severity of radiation dermatitis.

SECONDARY OUTCOMES:
Onset of radiation dermatitis | From radiotherapy start, until to 4 weeks post radiation therapy; up to 3 months
  Timepoint of onset of CTCAE v4.0 radiation dermatitis Grades 2 and/or 3 during or after radiotherapy.
Length of time until resolution of radiation dermatitis | From onset of radiation dermatitis, until radiation dermatitis resolution, up to 3 months
  Length of time from peak incidence to resolution of radiation dermatitis.
Patient reported symptoms treatment | From onset of radiation dermatitis, until radiation dermatitis resolution, up to 3 months
  Patient reported comfort scale obtained using the eviQ RISRAS form.
Cost-effectiveness | From radiotherapy start, until to 4 weeks post radiation therapy; up to 3 months
  The mean total cost of skin care per patient.
Incidence of late-effects skin toxicity | 3 - 12 months post radiation treatment
  The late skin toxicity post-radiotherapy assessed using the Radiation Therapy Oncology Group (RTOG) grading definitions:
  Grade 0: No change over baseline Grade I: Follicular, faint or dull erythema, epilation, dry desquamation, decreased sweating Grade II: Tender or bright erythema, patchy moist desquamation, moderate oedema Grade III: Confluent, moist desquamation other than skin folds, pitting oedema Grade IV: Ulceration haemorrhage, necrosis

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Townsville Cancer Center, Townsville Hospital and Health Service, Douglas, Queensland
  - Princess Alexandra Hospital, South Brisbane, Queensland